CLINICAL TRIAL: NCT03957629
Title: An Open, Multi-center Clinical Study of Combination Therapy With Tenofovir Disoproxil Fumarate and Peginterferon Alpha 2a in Nucleos(t)Ide Analogs Experienced Patients With HBV Related Hepatic Fibrosis.
Brief Title: Optimized Treatment of Peginterferon Alfa 2a in Treatment Experienced Patients With HBV Related Liver Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PL7
Record Dates: First submitted 2019-05-19; First posted 2019-05-21 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis B; Liver Fibrosis
Keywords: hepatitis b virus; liver fibrosis; peg interferon alfa-2a; tenofovir disoproxil fumarate
MeSH Terms: conditions — Hepatitis B; Liver Cirrhosis | interventions — Tenofovir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TDF group (Active Comparator): 93 patients would receive treatment of oral medication of tenofovir disoproxil fumarate (TDF) 300mg once per day from baseline to 48 weeks. Then they would receive oral medication of TDF 300 mg once per day from 49 to 96 weeks.
  Interventions: Drug: Tenofovir Disoproxil Fumarate
- Combination group (Active Comparator): 93 patients would receive treatment of subcutaneous injection of peginterferon alfa 2a 180 μg once per week and meanwhile oral medication of tenofovir disoproxil fumarate (TDF) 300 mg once per day from baseline to 48 weeks. Then they would receive oral medication of TDF 300 mg once per day from 49 to 96 weeks.
  Interventions: Drug: Tenofovir Disoproxil Fumarate; Drug: PEG-Interferon alfa 2a

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate — Oral medication of Tenofovir Disoproxil Fumarate 300mg once per day.
  Other Names: Viread; Beixin
Drug: PEG-Interferon alfa 2a — Subcutaneous injection of Peginterferon Alfa-2a 180 μg once per week.
  Other Names: Pegasys
  Arms: Combination group

SUMMARY:
Compared to TDF, peginterferon alfa 2a may has more therapeutic efficacy in hepatitis B surface antigen or e antigen seroconversion and anti-tumor occurrence in chronic hepatitis b patients. We design this study to compare the effectiveness and safety between the combination therapy of TDF and peg-IFN with TDF alone in NAs experienced patients with HBV related liver fibrosis. Especially the improvement of liver fibrosis and the occurrence of long-term end-stage liver disease such as cirrhosis, liver cancer, etc.

DETAILED DESCRIPTION:
Compared to TDF, peginterferon alfa 2a may has more therapeutic efficacy in hepatitis B surface antigen or e antigen seroconversion and anti-tumor occurrence in chronic hepatitis b patients. We design this study to compare the effectiveness and safety between the combination therapy of TDF and peg-IFN with TDF alone in NAs experienced patients with HBV related liver fibrosis. Especially the improvement of liver fibrosis and the occurrence of long-term end-stage liver disease such as cirrhosis, liver cancer, etc.

Main purpose: Comparing the improvement rate of liver fibrosis. Secondary purpose: Comparing the incidence of adverse events. Comparing the incidence of cirrhosis, hepatocellular carcinoma, and liver failure.

Comparing the rates of HBsAg and HBeAg serological conversion.

ELIGIBILITY:
Inclusion Criteria:

1. Positive hepatitis b surface antigen or hepatitis b virus DNA > 0.5 year;
2. Receiving treatment of nucleoside/nucleotide analogues at least one year before recruited;
3. Age from 18 to 55 years old;
4. Normal liver function(ALT<ULN,AST<ULN and TBil<ULN).
5. Undetectable hepatitis b virus DNA or less than 100IU/ml.
6. LSM between 6 and 12 kpa measured by fibroscan;
7. Liver ultrasound: normal or echo thickening, and portal vein diameter ≤ 12mm.

Exclusion Criteria:

1. Decompensated cirrhosis, hepatocellular carcinoma or other malignancy;
2. Pregnancy, lactation or female has plan of pregnancy within 18 months;
3. Accompanied with other active liver diseases(HAV, HCV, HDV, HEV, autoimmune liver disease, drug-induced liver injury, alcoholic liver disease, genetic metabolic liver disease, etc.)；
4. Accompanied with human immunodeficiency virus infection or congenital immune deficiency diseases;
5. Accompanied with severe diabetes, autoimmune diseases etc. and other important organ dysfunctions;
6. Patients who fail to comply with this research arrangement and sign an informed consent form
7. Patients can not follow-up;
8. Investigator considering inappropriate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Ratio of regression of fibrosis | 48 weeks; 96 weeks
  Regression of fibrosis was defined as liver stiffness measured by transient elastography changed from 9~12kpa to 6~9kpa or below, and from 6~9kpa to less than 6kpa. After treatment, the proportion of patients with regression of fibrosis in the two groups was the ratio of regression of fibrosis, separately.

SECONDARY OUTCOMES:
Ratio of loss of hepatitis b e antigen or/and seroconversion | 24 week, 48 week, 72 week, 96 week
  Hepatitis b e antigen and hepatitis b e antibody would be tested to know the ratio of patients with negative hepatitis B e antigen and positive hepatitis B e antibody at 4 time points after anti-virus treatment.
Ratio of loss of hepatitis b s antigen or/and seroconversion | 24 week, 48 week, 72 week, 96 week
  Hepatitis b s antigen and hepatitis b s antibody would be tested to know the ratio of patients with negative hepatitis B s antigen and positive hepatitis B s antibody at 4 time points after anti-virus treatment.
Logarithmic mean of HBsAg decline | 24 week, 48 week, 72 week, 96 week
  Hepatitis b s antigen would be tested to know the decline of patients with positive hepatitis B s antigen at 4 time points after anti-virus treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peng, ph.D., Study Director — Third Affiliated Hospital, Sun Yat-Sen University; Xu, ph.D., Study Director — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No